CLINICAL TRIAL: NCT01718613
Title: Vasopressin Versus Norepinephrine for the Management of Septic Shock in Cancer Patients
Acronym: VANCS II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Cristiane Maciel Zambolim, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP 1079/17
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Vasopressins; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Norepinephrine (Active Comparator)
  Interventions: Drug: Norepinephrine
- Vasopressin (Active Comparator)
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — Blinded Vasopressin will be started if there is persistent hypotension, characterized by mean arterial pressure <65 mmHg after fluid replacement
  Arms: Vasopressin
Drug: Norepinephrine — Blinded Norepinephrine will be started if there is persistent hypotension, characterized by mean arterial pressure <65 mmHg after fluid replacement
  Arms: Norepinephrine

SUMMARY:
Although arginine vasopressin has been used as an additional drug in refractory shock in worldwide clinical practice, there are no prospective studies using it as a first choice therapy in patients with cancer and septic shock.

The aim of this study is assess if the use of arginine vasopressin would be more effective on treatment of septic shock in cancer patients than norepinephrine, decreasing the composite end point of mortality and organ failure in 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Solid neoplasm needing ICU
* Septic Shock according standard criteria

Exclusion Criteria:

* Younger than 18 years;
* Pregnancy;
* Raynaud's phenomenon, systemic sclerosis or vasospastic diathesis;
* Severe hyponatremia (Na<130mEq/L);
* Acute mesenteric ischemia;
* Acute myocardial infarction;
* Cardiogenic shock;
* Current use of vasopressor before randomization
* Expected ICU stay less than 24 hours
* Enrolled in another study;
* Refusal to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28-day from randomization
  Mortality from all causes in 28-day follow-up

SECONDARY OUTCOMES:
90-days mortality | 90 days after randomization
  Mortality from all causes 90 days after randomization
Days alive and free of mechanical ventilation | 28 days after randomization
  Days alive and free of mechanical ventilation at 28-day follow-up
Days alive and free of vasopressors | 28 days after randomization
  Days alive and free of any type of vasopressor agent at 28-day follow-up
Days alive and free of renal replacement therapy | 28 days after randomization
  requirement of dialysis of hemofiltration at 28-day follow-up
SOFA score in 24 hours | 24 hours after ICU admission
  Severity of organ failure according to the Sequential Organ Failure Assessment (SOFA) score during the first 24 hours after randomization.
SOFA score in 96 hours | 96 hours after randomization
  Severity of organ failure according to the Sequential Organ Failure Assessment (SOFA) score during the first 96 hours after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane M Zambolim, MD, Principal Investigator — Department of Anesthesia and Critical Care, Intensive Care Unit - ICESP
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, Sao Paulo/SP, Brazil

REFERENCES:
- [Derived] Hajjar LA, Zambolim C, Belletti A, de Almeida JP, Gordon AC, Oliveira G, Park CHL, Fukushima JT, Rizk SI, Szeles TF, Dos Santos Neto NC, Filho RK, Galas FRBG, Landoni G. Vasopressin Versus Norepinephrine for the Management of Septic Shock in Cancer Patients: The VANCS II Randomized Clinical Trial. Crit Care Med. 2019 Dec;47(12):1743-1750. doi: 10.1097/CCM.0000000000004023. PMID 31609774